CLINICAL TRIAL: NCT02006225
Title: GCSF Plus Plerixafor as First-line Treatment for Autologous Stem Cells Harvest in Children With Malignant Diseases in Need for High-dose Chemotherapy With Stem Cell Rescue.
Brief Title: Stem Cell Harvesting Using GCSF Plus Plerxiafor, in First -Line, for Heavily Pre- Treated Pediatric Oncology Patients.
Acronym: GCSF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-13-MB-0693-12-CTIL
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-04

CONDITIONS: Autologous Stem Cell Transplantation
Keywords: autologous; stem cell; transplantation
MeSH Terms: interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plerixafor (Experimental): The use of plerixafor as additive measurment for the conventional stem cell collection protocol.
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor

SUMMARY:
Plerixafor has been intensively used in recent years for harvesting autologous stem cells from lymphoma and myeloma adult patients. Its use is indicated after failure to harvest with GCSF alone. Nevertheless, in the pediatric population its appliance is less well established and the indications are less well confirmed .Several disease states and diagnoses may prompt the anticipation of difficulties in harvesting stem cells using GCSF only. Such patients may benefit utilizing plerixafor in first-line rather than exhausting the stem cell niche with GCSF alone and only than go for plerixafor as second-line rescue procedure.

In this study we propose to examine the applicability and feasibility of harvesting autologous stem cells by means of GCSF + plerixafor in first-line measure for pediatric patients with specific indications.

DETAILED DESCRIPTION:
Improve and report outcomes of children undergoing peripheral stem and progenitor cell harvesting applying plerixafor in first-line aphaeresis, including:

Pre-harvesting FACS-derived CD34+ cell number. Number of stem cells harvested. Number of T-cells harvested. Days of hospitalization.

Procedure related toxicity including:

Infections. Line complications. Other organ toxicities.

Compare outcomes of plerixafor-derived stem and progenitor cells harvesting between different pediatric oncological diseases, including high-risk neuroblastoma, high-risk brain tumors, high-risk sarcomas and relapsed lymphomas.

Outcomes to be analyzed:

1. Peripheral blood stem cell content by means of percentage of CD34+ cells, after conditioning protocol (4 days of 10mcg/kg GCSF per day and one dose of plerixafor 0.24mg/kg 10 hours before collection) and before harvesting.
2. Number of stem cells harvested.
3. Morbidity:

   1. Bleeding at the time of catheter placement, during harvesting procedure and post harvesting.
   2. Infections: localized vs. generalized. Type of pathogen isolated.
4. Platelet number and hemoglobin level post harvesting.
5. kidney function.
6. Duration of hospitalization: Evaluation of the time course from the day of hospitalization for the harvesting to the day of discharge.

ELIGIBILITY:
Inclusion Criteria:

* The following patients will be included in this study:

Patients with high-risk neuroblastoma after third-line chemotherapy. Patients with high-risk medulloblastoma/PNET after spinal irradiation. Patients with primary sarcomas after third or more line therapies, Patients with relapsed lymphomas after third line chemotherapy. Patients with relapsed neuroblastoma, medulloblastoma, lymphoma or sarcoma after previous autologous stem cell transplantation.

Age equal to or less than 30 years at time of diagnosis. Patients eligible for AHCT according to their treating protocol or patients with neuroblastoma eligible for 131I-MIBG-therapy.

Patients with maligancies disease who candidates to autologous stem cell transplantation ,taking from them autologus stem cell as back up.

Exclusion Criteria:

Healthy stem cells donors

Patients who older than 30 years

Patients with non maligancies disease that candidates to autologous stem cell transplantation

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2019-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood stem cell content by means of percentage of CD34+ cells | After conditioning protocol (4 days of 10mcg/kg GCSF per day), and on the fifth day after one dose of plerixafor 0.24mg/kg, 10 hours before collection - before harvesting. After harvesting - the number of collected CD34+ cells.
  1. Peripheral blood stem cell content before harvesting by means of percentage of CD34+ cells, after conditioning protocol (4 days of 10mcg/kg GCSF per day) and after adding one dose of plerixafor 0.24mg/kg 10 hours before collection.
  2. Number of CD34+ stem cells that were collected after adding plerixafor with relation to the target number of stem cells needed.

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Bitan, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center